CLINICAL TRIAL: NCT04444102
Title: The Acute Impact of Yoga-based Stretching on Inflammation and Its Resolution: a Pilot Study
Brief Title: The Acute Impact of Yoga-based Stretching on Inflammation and Its Resolution
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Harvard University Faculty of Medicine (Other)
Responsible Party: Principal Investigator, Peter Wayne, Principal Investigator, Harvard University Faculty of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2019P001716
Record Dates: First submitted 2020-03-23; First posted 2020-06-23 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Inflammation; Fascia; Inflammation; Musculoskeletal Pain; Lower Back Pain; Neck Pain
Keywords: stretching; yoga; mind-body therapies; inflammation
MeSH Terms: conditions — Inflammation; Fasciitis; Musculoskeletal Pain; Low Back Pain; Neck Pain

STUDY DESIGN:
Intervention Model Description: The present study is a pilot randomized clinical trial (RCT) with 3 arms. These arms are: Control Group, Mild Stretching Group, and Intense Stretching Group. Ten participants will be allocated in each arm.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants and yoga-based stretching instructor are not blinded. Nurses and lab technicians are blinded during blood draws. Laboratory analysts are blinded during sample analyses. Statisticians will be unblinded once all laboratory analyses are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (CG) (No Intervention): Those subjects randomized to the CG will be offered reading options that do not evoke high emotional distress. They will spend an hour reading.
- Stretching protocol 1, Mild Stretching Group (MSG) (Experimental): The protocol starts with 5 minutes of instruction about finding a range of stretching representing approximately 50% of the range of motion and pain-free. The instructor will also wear wrist and ankle reflective bands as body-marks to show a posture with 100% stretch and then corrected to 50%. Once the participant grasps the concept the routine will begin with 5 minutes of warm-up, followed by stretching exercises targeting 10 anatomical groups. Each posture will last 1 minute divided in 30 seconds of settling into each posture and 30 seconds of holding. Each session will be video recorded to analyze the stretching range, only if the participant agrees at the informed consent visit. Participants will be encouraged to find their own 50% with some feedback from the instructor.
  Interventions: Procedure: Yoga-based stretching
- Stretching protocol 2, Intense Stretching Group (ISG): (Experimental): The protocol starts with 5 minutes of instruction about finding a range of stretching representing approximately 100% of the range of motion and pain-free. The instructor will also wear wrist and ankle reflective bands as body-marks to show a posture with 100% stretch. Once the participant grasps the concept the routine will begin with 5 minutes of warm-up, followed by stretching exercises targeting 10 anatomical groups. Each posture will last 1 minute divided in 30 seconds of settling into each posture and 30 seconds of holding. Each session will be video recorded to analyze the stretching range, only if the participant agrees at the informed consent visit. Participants will be encouraged to find their own 100% with some feedback from the instructor.
  Interventions: Procedure: Yoga-based stretching

INTERVENTIONS:
Procedure: Yoga-based stretching — Different yoga postures (ASANA) were isolated from conventional yoga practice to stretch different muscle groups.
  Muscle groups stretched: hip extensor and adductors, hip & plantar flexors, shoulder extensors, shoulder horizontal adductors, shoulder extensors-adductor, wrist flexor, trunk extensors, lateral flexors, and trunk rotators.
  Arms: Stretching protocol 1, Mild Stretching Group (MSG); Stretching protocol 2, Intense Stretching Group (ISG):

SUMMARY:
The goal of this study is to explore the impact of two types of yoga-based body stretching (mild and intense) on dynamic changes of Systemic Inflammatory Cytokines (SICs) and Specialized Pro-resolving Mediators (SPMs) in yoga-naïve subjects.

DETAILED DESCRIPTION:
During the last decade, yoga has become increasingly popular in Western cultures. The 2017 NIH report indicated that 14.3% of the adult population practice yoga in the USA. The most common yoga styles tested in randomized clinical trials (RCTs) are Hatha, Iyengar, and Patanjali.

One key physical component of yoga is the stretching that occurs during different postures. Based on animal studies, it is plausible to think that the physical intensity of stretching may affect systemic inflammatory outcomes, i.e. SICs and SPMs. However, human studies have not isolated and quantified the impact of stretching. In consequence, it is not known to what extent the benefits of yoga can be attributed to the physical aspect of stretching. One way to explore the effect of yoga would be to isolate the stretching element and compare two stretching protocols with yoga-based postures on SICs and SPMs.

In previous preclinical studies using an ex-vivo stretching model of mouse connective tissue (AICUC: 04996), the investigators found that fibroblasts are actively involved in the regulation of connective tissue tension, demonstrating that fibroblasts have a more elaborate scheme of responses to mechanical stress than was previously thought.

Later, in the inflammatory active stretch rat model (AICUC 04995), the investigators found that after 10 minutes of an active stretch there was a significant reduction in the inflammatory lesion size area measured with ultrasound and a reduction of infiltrating neutrophils. The SPM Resolvin 1 (RvD1) was also measured and showed a significant difference between the stretch and no stretch group. These promising results encouraged the investigators to keep exploring the fundamental innate mechanism by which the body enhances the healing of an inflammatory process regardless of its etiology; e.g., a mouse breast cancer model with active stretch showed that with four weeks of stretching once a day, tumors were reduced roughly to the half comparing with the no-stretch group and a pig study currently underway is exploring the effects of active stretching on SPMs production and determining changes in Polymorphonuclear Neutrophil (PMN) and macrophages migration toward the inflammatory stimulus.

These pre-clinical results motivated the research group to move forward with a translational pilot study to explore first the feasibility and second, the effect of stretching on the connective tissue and muscles of healthy humans. The investigators presume to find an effect of stretching on a systemic level. Hence, they propose to measure levels of SICs and SPMs, as well as their changes over time after one acute session of yoga-based stretching postures. The investigators plan to collect blood samples at baseline pre-intervention and then at 0 minutes, 30 minutes, 1, 2, and 3, and 24 hours after the intervention. Samples will be analyzed using flow cytometry and ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Age between 40 - 60 years old.
* Non-smoking
* BMI between 19 and 29.

Exclusion Criteria:

* Any history of chronic inflammatory disease or recent acute illness (< 1 month)
* Vaccination within the last 3 months
* Regular medication, or any medication in the preceding week
* Practice of structured higher-intensity exercise at least twice a week for more than 30 minutes
* Pregnancy
* Endocrine disorders (e.g. diabetes)
* Significant soft tissue injury
* Surgical supportive devices (nails, wire, screws, pins, plates) in an area of the body to be stretched (toes, ankles, knees, hips, shoulders, elbows, wrists, fingers and spine)
* Fractures in the past 3 years
* Generalized joint hypermobility or genetic conditions such as Marfan syndrome and Ehlers-Danlos syndrome
* Alcoholism (> 10 drinks per week) and drug abuse.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a pilot study including one session of acute stretching and serial blood samples over a period of 24 hours. | Two consecutive study visits per participants over a period of 24 hours
  * Study recruitment will be completed within 9 months
  * >70% of participants will complete two study visits
  * Participants will adhere to study protocol, including completion of outcome assessments (> 90%) and complying with stretching instructions specific to the mild and intense stretching protocol (confirmed with video analysis)
  * There will be no serious adverse events reported.

SECONDARY OUTCOMES:
Systemic inflammatory cytokines | Baseline, 0-, 30-, 60-, 120-, 180-minutes and 24 hours post intervention.
  Cytokines (IL-1b, IFN-a2, IFN-y, TNF-a, MCP-1, IL-6, IL-8, IL-10, IL-12p70, IL-17A, IL-18, IL-23, IL-33) Serum levels in pg/mL
Specialized pro-resolving mediators (SPMs) | Baseline, 0-, 30-, 60-, 120-, 180-minutes and 24 hours post intervention.
  Lipid mediators

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Wayne, PhD, Principal Investigator — Brigham and Women's Hospital and Harvard University
Locations (1):
- Ambulatory Clinical Center (ACC), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The results of this study may eventually be published, and information may be exchanged between medical investigators and collaborators, but patient confidentiality will be maintained. Institutional Review Board and regulatory authorities will be granted direct access to original medical and research records for verification of clinical trial procedures and/or data. If the record is used or disseminated for government purposes, it will be done under conditions that will protect the subject's privacy consistent with laws relating to public disclosure of information and the law-enforcement responsibilities of the agency (e.g. NIH and FDA).

REFERENCES:
- [Result] Ding D, Stamatakis E. Yoga practice in England 1997-2008: prevalence, temporal trends, and correlates of participation. BMC Res Notes. 2014 Mar 24;7:172. doi: 10.1186/1756-0500-7-172. PMID 24661723
- [Result] Tindle HA, Davis RB, Phillips RS, Eisenberg DM. Trends in use of complementary and alternative medicine by US adults: 1997-2002. Altern Ther Health Med. 2005 Jan-Feb;11(1):42-9. PMID 15712765
- [Result] Clarke TC, Barnes PM, Black LI, Stussman BJ, Nahin RL. Use of Yoga, Meditation, and Chiropractors Among U.S. Adults Aged 18 and Over. NCHS Data Brief. 2018 Nov;(325):1-8. PMID 30475686
- [Result] Kiecolt-Glaser JK, Bennett JM, Andridge R, Peng J, Shapiro CL, Malarkey WB, Emery CF, Layman R, Mrozek EE, Glaser R. Yoga's impact on inflammation, mood, and fatigue in breast cancer survivors: a randomized controlled trial. J Clin Oncol. 2014 Apr 1;32(10):1040-9. doi: 10.1200/JCO.2013.51.8860. Epub 2014 Jan 27. PMID 24470004
- [Result] Ospina MB, Bond K, Karkhaneh M, Tjosvold L, Vandermeer B, Liang Y, Bialy L, Hooton N, Buscemi N, Dryden DM, Klassen TP. Meditation practices for health: state of the research. Evid Rep Technol Assess (Full Rep). 2007 Jun;(155):1-263. PMID 17764203
- [Result] Ebnezar J, Nagarathna R, Yogitha B, Nagendra HR. Effect of integrated yoga therapy on pain, morning stiffness and anxiety in osteoarthritis of the knee joint: A randomized control study. Int J Yoga. 2012 Jan;5(1):28-36. doi: 10.4103/0973-6131.91708. PMID 22346063
- [Result] Langevin HM. Connective tissue: a body-wide signaling network? Med Hypotheses. 2006;66(6):1074-7. doi: 10.1016/j.mehy.2005.12.032. Epub 2006 Feb 17. PMID 16483726
- [Result] Benias PC, Wells RG, Sackey-Aboagye B, Klavan H, Reidy J, Buonocore D, Miranda M, Kornacki S, Wayne M, Carr-Locke DL, Theise ND. Structure and Distribution of an Unrecognized Interstitium in Human Tissues. Sci Rep. 2018 Mar 27;8(1):4947. doi: 10.1038/s41598-018-23062-6. PMID 29588511
- [Result] Wosczyna MN, Rando TA. A Muscle Stem Cell Support Group: Coordinated Cellular Responses in Muscle Regeneration. Dev Cell. 2018 Jul 16;46(2):135-143. doi: 10.1016/j.devcel.2018.06.018. PMID 30016618
- [Result] Levy BD, Clish CB, Schmidt B, Gronert K, Serhan CN. Lipid mediator class switching during acute inflammation: signals in resolution. Nat Immunol. 2001 Jul;2(7):612-9. doi: 10.1038/89759. PMID 11429545
- [Result] Serhan CN, Savill J. Resolution of inflammation: the beginning programs the end. Nat Immunol. 2005 Dec;6(12):1191-7. doi: 10.1038/ni1276. PMID 16369558
- [Result] Berrueta L, Muskaj I, Olenich S, Butler T, Badger GJ, Colas RA, Spite M, Serhan CN, Langevin HM. Stretching Impacts Inflammation Resolution in Connective Tissue. J Cell Physiol. 2016 Jul;231(7):1621-7. doi: 10.1002/jcp.25263. Epub 2015 Dec 10. PMID 26588184
- [Derived] Munoz-Vergara D, Schreiber KL, Langevin H, Yeh GY, Zhu Y, Rist P, Wayne PM. The Effects of a Single Bout of High- or Moderate-Intensity Yoga Exercise on Circulating Inflammatory Mediators: A Pilot Feasibility Study. Glob Adv Health Med. 2022 Dec 11;11:2164957X221145876. doi: 10.1177/2164957X221145876. eCollection 2022. PMID 36583069